CLINICAL TRIAL: NCT06407544
Title: Prospective Comparative Study Between Ultrasound-guided Quadratus Lumborum Block Versus Fascia Iliaca Compartment Block for Postoperative Pain and Cognitive Dysfunction Management in Patient Undergoing Hip Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hassan Ahmed Mohamed, assistant lecteurer anaethesia and ICU and pain management department sohag univerisity hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-04-07MD
Record Dates: First submitted 2024-05-02; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Pain and Cognitive Dysfunction Management in Hip Surgery
MeSH Terms: conditions — Pain | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (Q): (Active Comparator): including 20 patients with hip fractures will undergo ultrasound guided anterior QLB, will be administered 0.3 ml/kg of 0.125% bupivacaine (containing 1 mic/ml of dexmedetomidine and 5 mg of dexamethasone).
  Interventions: Procedure: peripheral nerve block; Drug: PCA device as rescue medication with IV morphine 1mg if VAS more than 4
- Group (F): (Active Comparator): including 20 patients with hip fractures will undergo ultrasound guided FIB, will be administered 0.3 ml/kg of 0.125% bupivacaine (containing 1 mic/ml of dexmedetomidine and 5 mg of dexamethasone).
  Interventions: Procedure: peripheral nerve block; Drug: PCA device as rescue medication with IV morphine 1mg if VAS more than 4
- Group (C): (Active Comparator): including 20 patients with hip fractures will receive ultrasound scanning for QLB or FIB with saline injection [26].
  Interventions: Procedure: peripheral nerve block; Drug: PCA device as rescue medication with IV morphine 1mg if VAS more than 4

INTERVENTIONS:
Procedure: peripheral nerve block — peripheral nerve block guided by ultra sound through Ultrasound-guided quadratus lumborum block versus FICB or fascia iliaca block
Drug: PCA device as rescue medication with IV morphine 1mg if VAS more than 4 — PCA device as rescue medication with IV morphine 1mg if VAS more than 4 with a 10 min lock-out time

SUMMARY:
Hip fractures are more common in older people due to osteoporosis. It is estimated that around six million patients worldwide will suffer hip fractures annually by 2050 as the population ages [1]. Clinically, hip surgery is a common and effective treatment for hip fractures. There will be an increasing number of older people undergoing hip surgery, including osteosynthesis and arthroplasty. However, severe surgical trauma, postoperative pain, and postoperative cognitive dysfunction (POCD) can be a considerable challenge for older people undergoing hip surgery [2, 3].The successful use of QLB with all approaches has been reported in case reports for the following surgical procedures: proctosigmoidectomy, hip surgery, above-knee amputation, abdominal hernia repair, breast reconstruction, colostomy, closure, radical nephrectomy, lower extremity vascular surgery, total hip arthroplasty, laparotomy, and colectomy.

Ultrasound-guided quadratus lumborum block (QLB) is a recently described fascial plane block in which the anesthetic is injected adjacently to the quadratus lumborum (QL) muscle with the goal of anesthetizing the nerves in the thoracolumbar region [17,18]. As a trunk nerve block, quadratus lumborum block (QLB) has been widely used for postoperative analgesia in patients undergoing abdominal and lower limb surgeries [19].

QLB can provide adequate analgesia and reduce opioid requirements after hip surgery [20]FICB or fascia iliaca block (FIB), first proposed in 1989, is a means ofblocking the three principal lumbar plexus nerves of the thigh with a single injection of local anesthetic delivered immediately dorsal to the fascia iliaca [21,22]. Indications of FICB are surgical anesthesia to the lower extremity, management of cancer pain and pain owing to inflammatory conditions of the lumbar plexus, and amelioration of acute pain following trauma, fracture, and burn [23]. Fascia Iliaca Block (FIB), which is widely used for postoperative analgesia in hip surgery, is a nerve block technique with proven efficacy[24].

ELIGIBILITY:
Inclusion Criteria:

age > 65 years ASA 1 , ASA 2 Montreal Cognitive Assessment (MoCA) score ≥ 26 before surgery scheduled for hip surgery

Exclusion Criteria:

patient refusal History of chronic pain or daily use of analgesics History of psychiatric disorder or inability to understand the consent form or how to use a visual analog scale (VAS) for pain measurement inability to communicate appropriately Allergy to any required drugs alcohol abuse Local infection at the injection site contraindications to neuraxial anesthesia long-term use of antidepressants or narcotic analgesics

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
VAS score | 2 years
  measure pain intensity (0-10)with scores ranging from 0 (no pain) to 10 (the worst possible pain).
MOCA score | 2 years
  measure post operative cognitive dysfunctionThe MOCA scores including visuospatial ability, naming, short-term memory, attention, language, abstraction, delayed recall, and orientation. MoCA states ranges may be used to grade severity: 18-25 = mild cognitive impairment, 10-17= moderate cognitive impairment and less than 10= severe cognitive impairment.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dhanwal DK, Dennison EM, Harvey NC, Cooper C. Epidemiology of hip fracture: Worldwide geographic variation. Indian J Orthop. 2011 Jan;45(1):15-22. doi: 10.4103/0019-5413.73656. PMID 21221218
- [Background] Yucuma D, Riquelme I, Avellanal M. Painful Total Hip Arthroplasty: A Systematic Review and Proposal for an Algorithmic Management Approach. Pain Physician. 2021 May;24(3):193-201. PMID 33988938
- [Background] Uzoigwe CE, O'Leary L, Nduka J, Sharma D, Melling D, Simmons D, Barton S. Factors associated with delirium and cognitive decline following hip fracture surgery. Bone Joint J. 2020 Dec;102-B(12):1675-1681. doi: 10.1302/0301-620X.102B12.BJJ-2019-1537.R3. PMID 33249907
- [Background] Baeriswyl M, Kirkham KR, Kern C, Albrecht E. The Analgesic Efficacy of Ultrasound-Guided Transversus Abdominis Plane Block in Adult Patients: A Meta-Analysis. Anesth Analg. 2015 Dec;121(6):1640-54. doi: 10.1213/ANE.0000000000000967. PMID 26397443